CLINICAL TRIAL: NCT00962026
Title: A Phase I, Open-label, Safety Study of Anti-inflammatory Therapy With Rilonacept in Adolescents and Adults With Type 1 Diabetes Mellitus
Brief Title: Rilonacept in Diabetes Mellitus Type 1: Safety Study
Acronym: RID-A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Perrin C White, Director of Pediatric Endocrinology, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IL1T-AI-1022
Record Dates: First submitted 2009-08-04; First posted 2009-08-19 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Interleukin 1; Type 1 diabetes mellitus; Rilonacept; Arcalyst
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — rilonacept

ARMS (1):
- Rilonacept (Experimental)
  Interventions: Drug: Rilonacept

INTERVENTIONS:
Drug: Rilonacept — Rilonacept given subcutaneously, dose per package labeling, once weekly.
  Other Names: Arcalyst, IL-1 Trap

SUMMARY:
This study is being done to see if an investigational drug called rilonacept is safe to use in patients with type 1 diabetes, and if it can slow the loss of the body's ability to secrete insulin in patients who are still able to make a small amount of insulin.

ELIGIBILITY:
Inclusion Criteria:

* Within 5 years of diagnosis of type 1 diabetes
* Between the ages of 16 to 45 years
* Have at least one diabetes-related autoantibody present
* Have mean C-peptide level > 0.2 nmol/L on a mixed meal tolerance test
* Be taking insulin
* Complete written informed consent

Exclusion Criteria:

* Taking inhaled or oral steroids (for example Advair, Orapred)
* Have an active infection
* Have serologic evidence of HIV, Hepatitis C, Hepatitis C, or tuberculosis
* Have ongoing use of medications known to affect glucose tolerance
* Have a live vaccine 90 days prior to, or during this study
* Taking any other experimental medication within the past 28 days
* Have prior treatment with rilonacept
* Have any complicating medical issues or abnormal clinical laboratory blood counts or results that interfere with study conduct; history of malignancies
* Pregnant or lactating females
* Males and females unwilling to use an acceptable method of contraception for the duration of the study

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2011-02; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of infection in study participants | 7 months

SECONDARY OUTCOMES:
Incidence and severity of other adverse effects in study participants | 7 months
Changes in participants' sex steroids (testosterone/estradiol) | 7 months
Changes in participants' HbA1c levels, insulin doses, and beta cell preservation | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Perrin C White, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Children's Medical Center, Dallas, Texas, United States